CLINICAL TRIAL: NCT04164745
Title: Efficacy and Safety Study of Anlotinib With Pembrolizumab in Adults With Programmed Cell Death-Ligand 1 (PD-L1)-Positive Treatment-naïve Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Li Zhang, professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L037
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: NSCLC
MeSH Terms: interventions — anlotinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Anlotinib plus Pembrolizumab (Experimental)
  Interventions: Drug: Anlotinib, oral capsule; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Anlotinib, oral capsule — Participants receive Anlotinib 12 mg p.o, qd on Days 1-14 of each 3-week cycle until progressive disease or unacceptable toxicity plus pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years).
Biological: Pembrolizumab — Participants receive Anlotinib 12 mg p.o, qd on Days 1-14 of each 3-week cycle until progressive disease or unacceptable toxicity plus pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 administrations (up to approximately 2 years).

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Anlotinib (AL3818) combined with pembrolizumab (MK-3475) in treatment-naïve adults with no prior systemic therapy for advanced non-small cell lung cancer (NSCLC) whose tumors have a programmed cell death-ligand 1 (PD-L1) Tumor Proportion Score (TPS) greater than or equal to 1%.

The primary study hypotheses is that the combination of Anlotinib and pembrolizumab is superior to pembrolizumab alone(historical data) as assessed by Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).

ELIGIBILITY:
Inclusion Criteria:

1. volunteered to join the study, signed the informed consent, had good compliance and cooperated with the follow-up.
2. age: ≥18 years old.
3. Histologically or cytologically confirmed locally advanced NSCLC(not suitable for or refuse to do radical radiotherapy and chemotherapy)/advanced NSCLC, have not previously received systemic treatment for locally advanced or advanced NSCLC. The completion time of previous neoadjuvant / adjuvant treatment for recurrent subjects should be ≥ 6 months.
4. Negative in EGFR,ALK and ROS1(tumor tissue sample results).
5. Has tumor tissue that demonstrates PD-L1 expression in ≥1% of tumor cells (TPS≥1%) as assessed by immunohistochemistry (IHC) 22C3 pharmDx assay at a central laboratory.
6. Diagnosed with advanced or recurrent NSCLC through pathology, with measurable nidus(using RECIST 1.1).
7. Has a life expectancy of ≥3 months.
8. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Has adequate organ function:

   1. .HB≥90g/L;
   2. ANC≥1.5×109/L；
   3. PLT≥100×109/L；
   4. WBC≥4.0×109/L and ≤15×109/L;
   5. ALT and AST≤1.5×ULN(≤5×ULN in patients with liver metastases);
   6. ALP≤2.5×ULN;
   7. TBiL≤1.5×ULN;
   8. ALB≥30g/L;
   9. TSH≤ULN(If abnormal, T3 and T4 levels should be examined; If T3 and T4 levels are normal, they can be enrolled);
   10. Cr≤1.5×ULN，and CrCL≥60mL/min(Cockcroft-Gault).
10. The woman patients of childbearing age who must agree to take contraceptive methods (e.g. intrauterine device, contraceptive pill or condom) during the research and within another 4 months after it; who are not in the lactation period and examined as negative in blood serum test or urine pregnancy test within 7 days before the research; The man patients who must agree to take contraceptive methods during the research and within another 120 days after it.

Exclusion Criteria:

1. Has an active autoimmune disease that has required systemic treatment. Replacement therapy is not considered a form of systemic treatment and is allowed.
2. Is receiving systemic steroid therapy within 3 days before the first dose of study treatment.
3. Live vaccines were administered within 4 weeks or possibly during the study.
4. Gene test results of tissue or blood samples confirmed the existence of EGFR, ALK and ROS1 variants.
5. CT or MRI showed that the distance between the tumor focus and the large blood vessel was less than or equal to 5 mm, or there was a large local invasion Blood vessels, or central tumor with high risk of bleeding, or obvious cavitary or necrotic tumor of lung.
6. Has active central nervous system metastasis (subjects who have completed treatment 21 days before randomization and have stable symptoms can be enrolled, but they need to be confirmed by imaging evaluation as no active bleeding symptoms, and have stopped systemic agitation Hormone therapy: dosage > 10mg / day prednisone or other effective hormones.
7. Has received prior therapy with Anlotinib, anti-PD-1(L1) or anti-CTLA-4 agents.
8. Has a known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for ≥5 years since initiation of that therapy.
9. Has significant cardiovascular impairment, such as a history of congestive heart failure greater than New York Heart Association Class II, unstable angina, myocardial infarction within 12 months of the first dose of study treatment, or cardiac arrhythmia associated with hemodynamic instability.
10. Has uncontrolled blood pressure (defined as systolic pressure≥140 mm Hg or diastolic pressure≥90 mm Hg).

    Has had an allogeneic tissue/solid organ transplant.
11. Abnormal coagulation (INR > 1.5 or PT > ULN + 4S or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolysis or anticoagulation. Note: on the premise of INR ≤ 1.5, it is allowed to use low-dose heparin (daily dosage for adults is 6000-12000 U) or low-dose aspirin (daily dosage ≤ 100mg) for prevention purposes.
12. Has arterial/venous thrombosis within 6 months, such as cerebrovascular accidents (including temporary ischemic stoke), deevenous thrombosis, and pulmonary embolism.
13. Has had clinically significant hemoptysis within 3 months before the study (more than 50ml hemoptysis per day); or clinically significant bleeding symptoms or clear bleeding tendency (such as gastrointestinal bleeding, bleeding gastric ulcer, Gastrointestinal bleeding, hemorrhagic gastric ulcer, stool occult blood + + or above in baseline, or suffer from vasculitis, etc.
14. Urine routine indicates urine protein ≥ + +, or confirms 24-hour urine protein content ≥ 1.0g.
15. Has congenital or acquired immune deficiency (such as HIV infection), or active hepatitis.
16. Has uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.
17. Take major surgical treatments, open biopsy, or get overt traumatic injury within 28 days before enrollment.
18. Has a previous and current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severe impairment of lung function, etc.
19. Has received allogeneic cell / tissue / organ transplantation.
20. According to the judgment of the researcher, there are other factors that may cause the study to be forced to terminate halfway, For example, other serious diseases (including mental diseases) need to be treated in combination, with serious laboratory abnormalities, and Court or social factors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2019-11-16 (Estimated); Primary Completion 2021-11-16 (Estimated); Study Completion 2022-11-16 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) as assessed by RECIST 1.1 | Up to approximately 24 months
  PFS is defined as the time from date of enrollment to the date of the first documentation of progressive disease (PD) or death from any cause, whichever occurs first per RECIST 1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as assessed by RECIST 1.1 | Up to approximately 24 months
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response(CR) or a Partial Response(PR) per RECIST 1.1.
Disease Control Rate (DCR) as assessed by RECIST 1.1 | Up to approximately 24 months
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or stable disease per RECIST 1.1.
Overall Survival (OS) | Up to 12 months after last patient last visit
  OS is defined as the time from date of enrollment to date of death from any cause.
Progression Free Survival 2 (PFS2) | Up to 12 months after last patient last visit
  PFS2 will be defined as beginning with enrollment and ending with the first of the following events: a) death; b) disease progression on any treatment given after 1st progression. The determination of disease progression will be based on RECIST 1.1 criteria.
Toxicity Rate | Up to 12 months after last patient last visit
  Toxicity Rate is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing adverse event (AE) including AE of all level, AE of grade 3/4, irAE

CONTACTS AND LOCATIONS:
Overall Officials: LI zhang, master, Principal Investigator — Peking Union Medical College Hospital, Beijing, China
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided